CLINICAL TRIAL: NCT04131231
Title: Safety and Effectiveness of Microparticles Packaging Chemotherapeutic Drugs(MPCD) Therapy on the Treatment of Malignant Pleural Effusion
Brief Title: Safety and Effectiveness of MPCD Therapy on the Treatment of Malignant Pleural Effusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Fei Ma, Deputy Director of Oncology Medicine, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC20180327
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer; Breast Cancer; Malignant Pleural Effusion
Keywords: microparticles packaging chemotherapeutic drugs; MPCD; malignant pleural effusion; MPE
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- microparticles packaging methotrexate (MPs-MTX) group (Experimental): Patients are first treated with microparticles packaging methotrexate (MPs-MTX) via intrapleural infusion four times on day5,6,7,8 and then undergo chemotherapy 1 cycle from day12. After 4 weeks from the beginning of the treatment (day1 of treatment), ORR is assessed.
  MPs-MTX: 5 U of MPs-MTX containing a total dose of more than 25μg of MTX dissolving in 50ml of physiological saline solution
  Interventions: Drug: microparticles packaging methotrexate (MPs-MTX)
- recombinant human interleukin-2(rhIL-2) group (Active Comparator): Patients are first treated with rhIL-2 via intrapleural infusion three times on day5,8,11 and then undergo chemotherapy 1 cycle from day12. After 4 weeks from the beginning of the treatment (day1 of treatment), ORR is assessed.
  rhIL-2: 2 million IU of rhIL-2 dissolving in 50ml of physiological saline solution
  Interventions: Drug: recombinant human interleukin-2(rhIL-2)

INTERVENTIONS:
Drug: microparticles packaging methotrexate (MPs-MTX) — 50ml, intrapleural infusion, day5,6,7,8
  Arms: microparticles packaging methotrexate (MPs-MTX) group
Drug: recombinant human interleukin-2(rhIL-2) — 50ml, intrapleural infusion, day5,8,11
  Arms: recombinant human interleukin-2(rhIL-2) group

SUMMARY:
This is a prospective, open-label , multicenter randomized controlled trial, with 248 cases in 50 centers planned for a period of 2 years. The aim of the study is to evaluate the safety and effectiveness of microparticles packaging chemotherapeutic drugs (MPCD) therapy on the treatment of malignant pleural effusion (MPE) in patients with advanced lung cancer or breast cancer.

DETAILED DESCRIPTION:
After obtaining informed consent, patients who meet the eligibility criteria will be randomly assigned 1:1 to treatment either with MPCD or recombinant human interleukin-2(rhIL-2) for injection. Randomization is stratified by tumor type and previous treatment. Patients in the MPCD group are first treated with microparticles packaging methotrexate (MPs-MTX) via intrapleural infusion four times on day5,6,7,8 and then undergo chemotherapy 1 cycle from day12. Patients in the control group are first treated with rhIL-2 via intrapleural infusion three times on day5,8,11 and then undergo chemotherapy 1 cycle from day12. After 4 weeks from the beginning of the treatment (day1 of treatment), the efficacy is assessed according to the WHO (1997) Response Evaluation Criteria In MPE and the evaluation methods mainly include physical examination, ultrasound and computed tomography (CT). The patients will be monitored by telephone every three months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed as lung cancer or breast cancer;
2. Cytologically or histologically confirmed MPE needing thoracocentesis treatment;
3. Without thoracocentesis treatment within 4 weeks;
4. ECOG PS score: 0-2 points;
5. Predicted life expectancy greater than 3 months;
6. 18 years ≤Age ≤80 years；
7. Bone marrow function: hemoglobin(HGB) ≥90g/L，white blood cells(WBC) ≥3.0×10^9/L，absolute neutrophil count(ANC) ≥1.5×10^9/L，platelets (PLT) ≥80×10^9/L，international standardized ratio (INR) <1.5;
8. Hepatic function：alanine aminotransferase(ALT) and aspartate aminotransferase(AST) ≤2.5×ULN，serum total bilirubin≤1.5× ULN;
9. Renal function：blood urea nitrogen(BUN) and serum creatinine(Cr) ≤1.5×ULN, or endogenous creatinine clearance rate(Ccr) ≥60mL/min;
10. Without other severe cardiac disease or respiratory disease;
11. The volunteers voluntarily join the study, sign informed consent, and have good compliance and follow-up.

Exclusion Criteria:

1. Inappropriate to receive chemotherapy;
2. Women who are pregnant, preparing to be pregnant, breastfeeding;
3. Known or suspected hypersusceptibility to any agents used in the treatment protocol;
4. With severe cardiac disease, respiratory disease, liver disease, kidney disease, or diabetes;
5. With severe infection;
6. With severe encapsulated pleural effusion or intrathoracic tissue adhesion which is inappropriate to receive thoracocentesis;
7. With cognitive impairment or low compliance;
8. Participating in other clinical trials within 4 weeks;
9. Undergoing immunotherapy within 3 months;
10. Other conditions considered to be inappropriate to be enrolled by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | 4 weeks
  Percentage of patients whose pleural effusion completely recover or reduce by more than 50% for more than 4 weeks

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 20 months
  Time from the date of first receive treatment to the date of first documented progression or date of death from any cause whichever came first
Overall Survival(OS) | up to 20 months
  Time from the date of first receive treatment to the date of death
Level of tumor markers | up to 20 months
  The change of the level of tumor markers(CEA,CA125) in blood and pleural effusion before and after treatment
Index of pleural effusion | up to 20 months
  Routine, biochemistry and cytological examination of pleural effusion

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, MD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science

IPD SHARING:
Plan to Share IPD: Undecided